CLINICAL TRIAL: NCT01514851
Title: Phase III Double-blind Comparative Study of BAY 77 1931 (Lanthanum Carbonate) With a Calcium Carbonate in Patients With Hyperphosphatemia Undergoing Hemodialysis
Brief Title: Phase III Double-blind Comparative Study of BAY77-1931 (Lanthanum Carbonate) With Calcium Carbonate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head Medical Development Japan, Bayer Yakuhin Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11877
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Hyperphosphatemia
Keywords: Hyperphosphatemia in ESRD (End Stage Renal Disease) patients on dialysis
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic | interventions — lanthanum carbonate; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): 750-2250mg/day, tid (three times a day), 8 weeks
  Interventions: Drug: Lanthanum carbonate (BAY77-1931)
- Arm 2 (Active Comparator): 1500-4500mg/day, tid, 8 weeks
  Interventions: Drug: Calcium carbonate

INTERVENTIONS:
Drug: Lanthanum carbonate (BAY77-1931)
  Arms: Arm 1
Drug: Calcium carbonate
  Arms: Arm 2

SUMMARY:
To assess the effect on reduction of serum phosphate and the safety of BAY77-1931 (Lanthanum Carbonate) in patients with hyperphosphatemia undergoing hemodialysis in a randomized, double-blind, parallel group study in comparison with Calcium carbonate.

ELIGIBILITY:
Inclusion Criteria:

* Pre-dialysis serum phosphate levels: ≧5.6 mg/dL and <11.0 mg/dL at 1 week after the initiation of the washout period.
* Out-patient
* Undergoing hemodialysis three times per week for at least previous 3 consecutive months

Exclusion Criteria:

* Pre-dialysis serum phosphate levels of ≧10.0 mg/dL at the start of the washout period or ≧11.0 mg/dL at 1 week after
* Corrected serum calcium level of <7.0 mg/dL or ≧11.0 mg/dL at the start of the washout period and/or 1 week after
* Serum intact PTH (Parathyroid) of ≧1000 pg/mL at the start of the washout period
* Pregnant woman, or lactating mother
* Significant gastrointestinal disorders including known acute peptic ulcer
* Liver dysfunction
* History of cardiovascular or cerebrovascular diseases
* Requiring treatment for hypothyroidism

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2006-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pre-dialysis serum phosphate levels (PSPL) at the end of the double-blind period | baseline to week 8
Presence/absence of incidence of hypercalcemia up to 8 weeks | up to 8 weeks

SECONDARY OUTCOMES:
Number of participants achieving target PSPL and time to achievement | up to 8 weeks
Serum calcium x phosphate product at the end of the double-blind treatment period | Week 8
Serum intact-PTH (Parathyroid) levels | Week 8
Serum calcium level corrected by serum albumin level at the end of the double-blind treatment period | Week 8
Number of participants achieving the target serum calcium levels | Week 8
Safety variables will be summarized using descriptive statistics based on adverse events collection | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (28):
- Japan (28):
  - Toyohashi, Aichi-ken
  - Yatomi, Aichi-ken
  - Asahi, Chiba
  - Chiba, Chiba
  - Kashiwa, Chiba
  - Matsudo, Chiba
  - Narita, Chiba
  - Kurume, Fukuoka
  - Isesaki, Gunma
  - Hiroshima, Hiroshima
  - Kobe, Hyōgo
  - Mito, Ibaraki
  - Tsuchiura, Ibaraki
  - Takamatsu, Kagawa-ken
  - Kochi, Kochi
  - Ōsaki, Miyagi
  - Sendai, Miyagi
  - Okayama, Okayama-ken
  - Suita, Osaka
  - Saitama, Saitama
  - Fuji, Shizuoka
  - Hamamatsu, Shizuoka
  - Tokushima, Tokushima
  - Arakawa-ku, Tokyo
  - Kodaira, Tokyo
  - Nerima-ku, Tokyo
  - Shibuya-ku, Tokyo
  - Shinjyuku-ku, Tokyo